CLINICAL TRIAL: NCT01671020
Title: Open-label, Randomized, Crossover Clinical Trials for Single Oral Dose of 60mg Fimasartan and Single IV Infusion of 30mg Fimasartan to Evaluate the Absolute Bioavailability of Kanarb® Tablet (Fimasartan) in Healthy Subjects
Brief Title: Clinical Trials for Single Oral Dose of 60mg Fimasartan and Single IV Infusion of 30mg Fimasartan to Evaluate the Absolute Bioavailability of Kanarb® Tablet (Fimasartan) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A657-BR-CT-115
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: fimasartan; absolute bioavailability
MeSH Terms: interventions — fimasartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (R)(T) (Active Comparator): Period 1: Fimasartan 60mg → Period 2: Fimasartan 30mg
  Interventions: Drug: Fimasartan
- (T)(R) (Active Comparator): Period 1: Fimasartan 30mg → Period 2: Fimasartan 60mg
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Fimasartan — Period 1 fisrt administration of fimasartan 60mg Period 2 second administration of fimasartan 30mg
  Arms: (R)(T)
Drug: Fimasartan — Period 1 first administration of fimasartan 30mg Period 2 second administration of fimasartan 60mg
  Arms: (T)(R)

SUMMARY:
Open-label, randomized, crossover clinical trials for single oral dose of 60mg fimasartan and single IV infusion of 30mg fimasartan to evaluate the absolute bioavailability of Kanarb® tablet (fimasartan) in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 55 years
* body weight: standard weight(Broca's index, Possible range is plus or minus 20percent)
* written informed consent

Exclusion Criteria:

* known allergy to Fimasartan
* existing cardiac or hematological diseases
* existing hepatic and renal diseases
* existing gastrointestinal diseases
* acute or chronic diseases which could affect drug absorption or metabolism history of any serious psychological disorder
* abnormal diet which could affect drug absorption or metabolism
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* participation in a clinical trial during the last 90 days prior to the start of the study

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
AUCinf, AUC, Cmax, Tmax, half-life; t1/2z, AUCt, Vdss, Cl, | PO : 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48hr, IV : 0.25, 0.5, 0.75, 1, 1.08, 1.17, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48hr

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, M.D, Ph.d, Principal Investigator — Division of Clinical Pharmacology
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea